CLINICAL TRIAL: NCT00954720
Title: A Prospective Observational Study of Iron Overload in Patients With Acute Leukemia or Myelodysplastic Syndromes Undergoing Myeloablative Allogeneic Stem Cell Transplantation
Brief Title: Observational Study of Iron Overload in Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Philippe Armand, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 07-413
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome
Keywords: AML; ALL; MDS; iron overload
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Iron Overload

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Banked serum and mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient undergoing transplant: Patients with acute leukemia or MDS undergoing ablative stem cell transplantation. No intervention.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no intervention on this trial

SUMMARY:
Recent retrospective studies have suggested that iron overload is a clinically important problem in patients undergoing ablative stem cell transplantation. However, these studies relied on serum ferritin as a surrogate of iron overload, which limits the conclusions that can be drawn from such analyses. Therefore, the investigators are conducting a prospective study to more rigorously examine the prevalence, mechanisms, and consequences of iron overload in this patient population.

DETAILED DESCRIPTION:
As above.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically confirmed acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), or myelodysplastic syndrome (MDS)
* Planned allogeneic stem cell transplantation with myeloablative conditioning regimen (regardless of stem cell source or donor HLA match)
* Patients will be eligible even if they have had prior stem cell transplantation (autologous or allogeneic)

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (MRI):

  * Patients with cardiac pacemakers, implanted cardiac defibrillator (ICD), cardiac electrodes, pacing wires, internal electrodes, cochlear, otologic or other ear implants, metallic fragments or foreign body, metallic prosthesis. Patients with surgical staples should not be imaged until 7 days post-op unless approved by a radiologist;
  * Severe claustrophobia
  * Note: a history of allergic reaction to gadolinium is not a contraindication to enrollment, as contrast will not be used.
* Inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient's who are 18 years or older with acute leukema or MDS underdoing a myeloablative allogeneic stem cell transplant
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2008-03; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To estimate the prevalence of pre-transplantation iron overload (defined as liver iron content >2 mg/g dry weight by MRI) and of pre-transplantation severe iron overload (defined as liver iron content >7 mg/g dry weight by MRI) | Pre-transplant

SECONDARY OUTCOMES:
To estimate the 6-month and 12-month prevalence of iron overload determined by liver MRI • To compare 6-month and 1-year TRM between patients with severe pre-transplantation iron overload (>7 mg/g dry weight) and those without. | 1 year post-transplant
To compare 6-month and 1-year TRM between patients with pre-transplantation serum ferritin > 2500 ng/ml and those with ferritin ≤ 2500 ng/ml. | 6 month and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Armand, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States